CLINICAL TRIAL: NCT00456417
Title: Evaluation of [123I] MNI-187 and SPECT as a Marker of Beta-amyloid Protein Deposition in Subjects With Alzheimer Disease in Comparison to Healthy Subjects
Brief Title: Evaluation of [123I] MNI-187 and SPECT in Patients With Alzheimers Disease in Comparison to Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institute for Neurodegenerative Disorders (Other)
Collaborators: Molecular NeuroImaging (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MNI-187-01
Expanded Access: Available
Record Dates: First submitted 2007-04-03; First posted 2007-04-05 (Estimated); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Alzheimers Disease
Keywords: Neurological; Alzheimers
MeSH Terms: conditions — Alzheimer Disease; Neurologic Manifestations | interventions — X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: 123-I MNI-187 Injection and Imaging Procedures

SUMMARY:
The underlying goal of this study is to assess 123-I MNI-187 SPECT imaging as a tool to detect ß-amyloid deposition in the brain of AD research participants and age- and gender-matched healthy subjects.

DETAILED DESCRIPTION:
Approximately 14 patients with Alzheimer's disease (AD) and 12 healthy controls will be recruited to participate in this study. Healthy controls will be examined to ensure that there is no evidence of neurodegenerative changes including cognitive decline.

All subjects will undergo written informed consent and a screening evaluation including baseline clinical laboratory testing, a baseline physical and neurological evaluation and baseline cognitive evaluations.

Subjects will be asked to undergo a bolus injection of 123-I MNI-187. Subjects will undergo serial SPECT imaging scans and serial venous plasma sampling for measurement of 123-I MNI-187 in plasma (both protein bound and free) over a period of up to 6 hours.

Subjects may be asked to undergo a second imaging visit between 2 and 6 weeks following the initial imaging visit following similar procedures to the initial imaging visit to evaluate the reproducibility of the imaging measure using this procedure. The imaging analyses will be performed by an image-processing specialist who will remain masked to the procedures employed with each imaging acquisition.

The primary imaging outcome measure will be the brain regional distribution volumes expressed as a brain tissue to plasma ratio of the radioligand, 123-I MNI-187. Time to the peak uptake and amplitude of the peak uptake will be evaluated for all brain regions and the results for the AD patients and controls will be compared.

For those subjects undergoing repeat imaging visits, the data from the initial scan will be compared to the second scan to determine which offers the reproducibility of the imaging outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* The participant is 50 years or older.
* Written informed consent is obtained.
* Participants have a clinical diagnosis of Alzheimer's disease based on National Institute of Neurological and Communicative Disorders and Stroke/Alzheimer's Disease and Related Disorders Association (NINCDS/ADRDA) criteria.
* Mini-Mental Status Exam score >16 and < 25.
* Modified Hachinski Ischemia Scale score of ≤ 4.
* Geriatric Depression Scales (GDS) ≤ 10.
* For females, non-child bearing potential or negative urine or blood pregnancy test on day of 123-I MNI-187 injection.

Exclusion Criteria:

* The subject has signs or symptoms of another neurodegenerative disease including Parkinson's disease, diffuse Lewy body dementia, or history of significant cerebrovascular disease.
* The subject has a clinically significant abnormal laboratory value and/or clinically significant unstable medical or psychiatric illness
* The subject has any disorder that may interfere with drug absorption distribution, metabolism, or excretion (including gastrointestinal surgery).
* The subject has evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, neurological, immunodeficiency, pulmonary, or other disorder or disease.
* Pregnancy

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-04; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
To assess the dynamic uptake and washout of 123-I MNI-187

SECONDARY OUTCOMES:
Blood metabolite characterization of 123-I MNI-187 in healthy and AD subjects to determine the metabolic fate and nature of metabolites; Evaluate the test/retest reproducibility of 123-I MNI-187 and SPECT in AD subjects and healthy controls | 1 yr

CONTACTS AND LOCATIONS:
Overall Officials: Danna Jennings, MD, Principal Investigator — Institute for Neurodegenerative Disorders
Locations (1):
- Institute for Neurodegenerative Disorders, New Haven, Connecticut, United States